CLINICAL TRIAL: NCT02381132
Title: A Randomized, Open Label, Prospective Study to Explore the Clinical Characteristics of Oral MNK155 and Norco 7.5mg/325 When Used for the Treatment of Moderate to Severe Post Operative Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Neil Singla (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor-Investigator, Neil Singla, Coordinating Investigator, Lotus Clinical Research, LLC
Organization: Lotus Clinical Research, LLC (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: LCR-MNK-155-01C
Record Dates: First submitted 2015-01-20; First posted 2015-03-06 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — oxycodone-acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MNK155 (Active Comparator): Hydrocodone Bitartrate/Acetaminophen Extended-Release Tablets
  Interventions: Drug: MNK155
- Norco 7.5mg/325mg (Active Comparator): Norco 7.5mg/325mg
  Interventions: Drug: Norco 7.5mg/325

INTERVENTIONS:
Drug: Norco 7.5mg/325
  Arms: Norco 7.5mg/325mg
Drug: MNK155
  Arms: MNK155

SUMMARY:
The purpose of this study is to explore the clinical characteristics oral MNK155 and Norco® 7.5mg/325mg when used for the treatment of moderate to severe post operative pain.

DETAILED DESCRIPTION:
This is a single center, open label, prospective, randomized study on adult post operative subjects who are expected to require oral opioid analgesia for at least 48 hours after surgery. The main study drug of interest in this study is MNK 155. Norco® 7.5mg/325mg is being utilized only as active comparator.

Subjects will be at least 18 years of age and will be scheduled to undergo elective surgery. The following surgical types will be allowed, although the list is not all inclusive:

* Abdominal surgery
* Soft tissue surgery
* Orthopedic surgery
* Spine surgery
* Genitourinary surgery

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who provide written informed consent prior to enrollment.
2. Male or female and 18 years of age or older.
3. Subjects who are scheduled to undergo elective general surgery including, but not limited to the following surgical types:

   * Abdominal surgery
   * Orthopedic surgery
   * Spine surgery
   * Genitourinary surgery
4. Subjects classified as American Society of Anesthesiologists (ASA class I-III).
5. Female subjects are eligible only if all of the following apply:

   * Not pregnant (subjects of child bearing potential must have a negative beta human chorionic gonadotropin (β-hCG) pregnancy test before surgery);
   * Not lactating;
   * Not planning to become pregnant within the duration of the study;
6. Subjects who are expected to have acute pain requiring oral opioid analgesics for at least 48 hours during the post operative period (either inpatient or outpatient).
7. Subjects who are willing and capable of understanding and cooperating with the requirements of the study.
8. Subjects able to understand and communicate in English.

Exclusion Criteria:

1. Subjects with a medical condition that, in the Investigator's opinion, could adversely impact the subject's participation, safety, or conduct of the study such as but not limited to a history of severe renal or hepatic impairment, severe active hepatic disease, or any other clinically significant medical condition that may preclude safe study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Post-operative Pain Control | 48 hours
  Patient Global Assessment

SECONDARY OUTCOMES:
Post-operative Pain Control | 120 hours
  Patient Global Assessment
Post-operative Pain Control as Assessed by the Healthcare Professional | 48 and 120 hours
  Healthcare Professional Global Assessments
Subject Satisfaction Regarding Ease of Use and Pill Burden | 48 hours and 120 hours after treatment initation
  Patient Satisfaction/Ease of Use and Pill Burden Assessment
Subject Reported Worst Pain (Secondary to Analgesic Gaps) | 24 hours after treatment initiation
  Assessment of Worst Pain- Numerical Rating Scale (NRS)
Total Daily Acetaminophen Exposure | 24 hours, 48 hours, 72 hours, 96 hours and 120 hours after treatment initation
  Number of Dosed of Acetaminophen
Sleep Disturbance | 24 hours, 48 hours and 72 hours after treatment initiation
  Assessment of Sleep Disturbance/Pain Interference with Sleep
Opioid Related Symptoms | 48 hours after treatment initiation
  Opioid Related Symptom Distress Scale (ORSDS)
Pill Diversion | Day 5
  Number of Pills Remaining and Accountability

CONTACTS AND LOCATIONS:
Locations (1):
- Lotus Clinical Research, LLC, Pasadena, California, United States